CLINICAL TRIAL: NCT02616445
Title: A Phase I Double-Blind, Randomised, Placebo-Controlled, Multiple Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of UE2343 in Healthy Subjects
Brief Title: Phase I MAD, Fed-Fasted, CSF Study of UE2343 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Actinogen Medical (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry); Linear Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: ACW0001
Record Dates: First submitted 2015-11-05; First posted 2015-11-30 (Estimated); Last update posted 2025-01-22 (Actual); Status verified 2017-05

CONDITIONS: Healthy Volunteers
Keywords: Xanamem; emestedastat
MeSH Terms: interventions — UE2343

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- MAD Study (Placebo Comparator)
  Interventions: Drug: UE2343; Drug: Placebo
- Fed-Fasted (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: UE2343
- CSF (Experimental)
  Interventions: Drug: UE2343

INTERVENTIONS:
Drug: UE2343 — * UE2343
  * 10mg, 20, 35mg
  * twice daily for 9 days
  Arms: MAD Study
Drug: Placebo — * 10mg, 20, 35mg
  * twice daily for 9 days
  Arms: MAD Study
Drug: Placebo — * Cross-over study
  * single dose administered twice (on day 1 and day 8)
  * study duration 17 days
  Arms: Fed-Fasted
Drug: UE2343 — * Cross-over study
  * UE2343
  * single dose administered twice (on day 1 and day 8)
  * study duration 17 days
  Arms: Fed-Fasted
Drug: UE2343 — * UE2343
  * twice daily for 3 days
  * single dose on day 4
  Arms: CSF

SUMMARY:
The purpose of this study is to determine whether the drug UE2343, a potential treatment for Alzheimer's Disease (AD), is effective by assessing safety, tolerability, pharmacokinetics and pharmacodynamics in a Multiple Ascending Dose Study. Protocol amendments to the study will examine any food effect and determine if the drug penetrates the Blood-Brain Barrier.

DETAILED DESCRIPTION:
Part 1 of this study is a double-blind, randomised, placebo-controlled, multiple ascending dose study to assess the safety, tolerability, PK and PD in healthy participants dosed twice daily at levels of 10, 20 and 35mg for 10 days.This part of the study will recruit 3 groups of 8 participants each.

Part 2 is a cross-over study to assess the effects of food on the PK of UE2343 in healthy participants dosed with two single doses at a level decided from Part 1. This part of the study will recruit a total of 12 participants.

Part 3 seeks to determine the PK of the UE2343 in CSF of healthy participants dosed twice daily for 4 days with a dose level determined from Part 1 and 2. This part of the study will recruit 4 participants.

Strategies to ensure adherence to the study include the requirement that participants remain at the clinical research facility for the duration of their participation in the study; drug accountability checks (i.e. reconciliation of used and unused capsules) by an independent clinical research associate; and administration of the capsules to the participant by a member of the study site team.

ELIGIBILITY:
Inclusion Criteria:

* Willing to use specified contraception
* BMI within specified range
* No clinically significant abnormalities in the results of laboratory evaluations at Screening and Day -1.

Exclusion Criteria:

* Abnormal medical history, including history of dementia
* No significant allergic reactions
* No prior drug or alcohol abuse
* Use of regular prescribed medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-02; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Assess Safety and Tolerability of UE2343 over 17 days including AEs, 12-lead ECGs, vital signs, Nerve conduction velocity, Labs. | Up to Day 17
Assess the Pharmacokinetic (PK) Plasma Parameter Maximum Plasma Concentration (Cmax) of UE2343 after a single dose | Day 1 and Day 8
Assess the Pharmacokinetic (PK) Plasma Parameter Time to Cmax (Tmax) of UE2343 after a single dose | Day 1 and Day 8
Assess the Pharmacokinetic (PK) Plasma Parameter Area Under the Curve (AUC) of UE2343 after a single dose | Day 1 and Day 8
Assess the Pharmacokinetic (PK) Plasma Parameter Terminal Elimination Half Life (t½) of UE2343 after a single dose | Day 1 and Day 8
Assess PK Parameter Maximum Plasma Concentration (Cmax) of UE2343 in CSF | Day 4

SECONDARY OUTCOMES:
Assess Pharmacokinetics (PK) Plasma parameter Maximum Plasma Concentration (Cmax) from time of dosing to 12 hours | Day 1 and Day 10
Assess Pharmacokinetics (PK) Plasma parameter Time to Cmax (Tmax) from time of dosing to 12 hours | Day 1 and Day 10
Assess Pharmacokinetics (PK) Plasma parameter Area Under the Curve (AUC) from time of dosing to 12 hours | Day 1 and Day 10
Assess Pharmacokinetics (PK) Plasma parameter Terminal Elimination Half Life (t½) from time of dosing to 12 hours | Day 1 and Day 10
Assess Pharmacokinetics (PK) Urine parameters (Amount of drug excreted in urine (Ae) and Ae as a % of dose) from time of dosing to 24 hours | Day 1 and Day 10
Assess PK Parameter Maximum Plasma Concentration (Cmax) of UE2343 in CSF compared to the Cmax value obtained in plasma | Day 4
Assess Pharmacodynamics (PD) Blood parameter Adrenocorticotropic hormone (ACTH) from baseline to end of study | Days 1, 10, 11, 12, 13 and 17.
Assess Pharmacodynamics (PD) Blood parameter Serum Cortisol from baseline to end of study | Days 1, 10, 11, 12, 13 and 17.
Assess Pharmacodynamics (PD) Blood parameter for Adrenal Androgens from baseline to end of study | Days 1, 10, 11, 12, 13 and 17.
Assess Pharmacodynamics (PD) Urine parameter Urinary Free Cortisol (UFF) from baseline to end of study | Days 1, 10, 11 and 12
Assess Pharmacodynamics (PD) Urine parameter Urinary Free Cortisone (UFE) from baseline to end of study | Days 1, 10, 11 and 12
Assess Pharmacodynamics (PD) Urine parameter 5α-tetrahydrocortisol (5αTHF) from baseline to end of study | Days 1, 10, 11 and 12
Assess Pharmacodynamics (PD) Urine parameter 5β-tetrahydrocortisol (5βTHF) from baseline to end of study | Days 1, 10, 11 and 12
Assess Pharmacodynamics (PD) Urine parameter tetrahydrocortisone (THE) from baseline to end of study | Days 1, 10, 11 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Ruffles, Study Chair — Actinogen Medical; Janakan Krishnarajah, Principal Investigator — Linear Clinical Research Limited
Locations (1):
- Linear Clinical Research, Nedlands, Western Australia, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Webster SP, McBride A, Binnie M, Sooy K, Seckl JR, Andrew R, Pallin TD, Hunt HJ, Perrior TR, Ruffles VS, Ketelbey JW, Boyd A, Walker BR. Selection and early clinical evaluation of the brain-penetrant 11beta-hydroxysteroid dehydrogenase type 1 (11beta-HSD1) inhibitor UE2343 (Xanamem). Br J Pharmacol. 2017 Mar;174(5):396-408. doi: 10.1111/bph.13699. Epub 2017 Jan 25. PMID 28012176